CLINICAL TRIAL: NCT05256979
Title: Clinical Observation of the Effect of Ursodeoxycholic Acid on Parameters Affecting Liver, Metabolic and Cardiovascular Morbidity and Mortality - Pilot Project
Brief Title: Ursodeoxycholic Acid in Patients With NAFLD - Clinical Observation
Acronym: URSO
Status: Active, not recruiting | Type: Observational
Sponsor: General University Hospital, Prague (Other)
Responsible Party: Principal Investigator, Radan Bruha, Principal Investigator, General University Hospital, Prague
Other Study IDs: GUHPrague
Record Dates: First submitted 2022-02-08; First posted 2022-02-25 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Non-Alcoholic Fatty Liver Disease
Keywords: NAFLD; Liver steatosis; Liver fibrosis; Ursodeoxycholic acid
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients with NAFLD indicated for ursodeoxycholic acid treatment ("by SPC: cholestatic hepatitis") will be offered an observational study. Examinations will be performed before the treatment and after 6month period. Laboratory parameters, non-invasive indices, liver elastography, cardiovascular parameters and liver MR spectroscopy will be performed.

DETAILED DESCRIPTION:
Patients with NAFLD newly indicated for ursodeoxycholic acid treatment will be offered an observational study. Clinical examinations, blood sampling, ultrasound examinations of the liver and liver elastography will be performed. Non-invasive indices evaluating liver fibrosis and steatosis based on common anthropometric and laboratory parameters (FLI, NAFLD fibrosis score, BARD score, APRI, FIB-4) will also be evaluated. The examinations will be repeated after 6 months of treatment (all as part of regular routine check-ups performed in patients with NAFLD). Before and after the follow-up, patients will be offered examinations as part of cardiovascular disease (ultrasound examination of the carotid artery and endothelial dysfunction) and examinations for quantification of hepatic steatosis by MR spectroscopy.

Statistical processing: individual parameters will be evaluated before the start of monitoring and after 6-month monitoring. A difference of p≤0.05 will be considered a statistically significant change.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with NAFLD with ALT elevation and cholestatic features who are indicated for standard treatment with ursodeoxycholic acid according to SPC ("Hepatitis of various etiologies with cholestatic syndrome").

Exclusion Criteria:

* Previous treatment with ursodeoxycholic acid.
* Diagnosis of cirrhosis at the start of the study.
* Etiology of liver disease other than NAFLD.
* Presence of malignant disease.
* Cardiovascular comorbidity: CHD / CHD on pharmacological therapy, history of myocardial infarction, stroke and coronary / carotid intervention.
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with NAFLD
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-07-02 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
The effect of urso on GGT | 6 months
  The effect of UDCA therapy on GGT activity (ukat/l; change from baseline).
The effect of urso on liver fat content | 6 months
  The effect of UDCA therapy on liver fat content measured by MR spectroscopy (percentual change from baseline).
The effect of urso on cardiovascular parameters - carotid intima media | 6 months
  The effect of UDCA therapy on carotid intima media thickness measured by ultrasound (change in mm from the baseline)
The effect of urso on cardiovascular parameters - endothelial dysfunction | 6 months
  The effect of UDCA therapy on endothelial dysfunction measured in percentual change in ENDO-PAT examination.

OTHER OUTCOMES:
The effect of urso on bile acid metabolism | 6 months
  To assess the effect of UDCA therapy on bile acid metabolism measured as percentual change in blood from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Radan BRUHA, Prof., Principal Investigator — General University Hospital, Prague
Locations (1):
- General University Hospital, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Vitek L. Bile Acids in the Treatment of Cardiometabolic Diseases. Ann Hepatol. 2017 Nov;16(Suppl. 1: s3-105.):s43-s52. doi: 10.5604/01.3001.0010.5496. PMID 29080341
- [Background] Sanchez-Garcia A, Sahebkar A, Simental-Mendia M, Simental-Mendia LE. Effect of ursodeoxycholic acid on glycemic markers: A systematic review and meta-analysis of clinical trials. Pharmacol Res. 2018 Sep;135:144-149. doi: 10.1016/j.phrs.2018.08.008. Epub 2018 Aug 9. PMID 30099154
- [Result] Ratziu V, de Ledinghen V, Oberti F, Mathurin P, Wartelle-Bladou C, Renou C, Sogni P, Maynard M, Larrey D, Serfaty L, Bonnefont-Rousselot D, Bastard JP, Riviere M, Spenard J; FRESGUN. A randomized controlled trial of high-dose ursodesoxycholic acid for nonalcoholic steatohepatitis. J Hepatol. 2011 May;54(5):1011-9. doi: 10.1016/j.jhep.2010.08.030. Epub 2010 Oct 31. PMID 21145828
- [Result] Ampuero J, Gallego-Duran R, Romero-Gomez M. Association of NAFLD with subclinical atherosclerosis and coronary-artery disease: meta-analysis. Rev Esp Enferm Dig. 2015 Jan;107(1):10-6. PMID 25603326